CLINICAL TRIAL: NCT05393492
Title: Dialectical Behavior Therapy for Challenging Behaviors and Emotional Distress After Acquired Brain Injury : a Pilot Study
Brief Title: Regulating Emotions and Behaviors After Brain Injury
Acronym: GREMO-LCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8264
Record Dates: First submitted 2022-01-18; First posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Acquired Brain Injury; Stroke/ Cerebrovascular Accident (Ischemic or Hemorrhagic); Brain Tumor (After Recovery); Encephalitis; Cerebral Anoxia; Meningitis
Keywords: brain injury; dialectical behavior therapy; emotions; emotional dysregulation; behavioral disorders; spirituality; challenging behaviors; linguistic markers; emotional distress; family burden; free will; interpretative phenomenological analysis; single-case experimental design
MeSH Terms: conditions — Brain Injuries; Stroke; Ischemia; Brain Neoplasms; Encephalitis; Hypoxia, Brain; Meningitis; Mental Disorders | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Intervention Model Description: DBT for patients
Who Masked: Outcomes Assessor
Masking Description: Blinded analysis of linguistic markers of emotional regulation and free will by an independent laboratory
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GREMO patients (Experimental): 1. 5 months of baseline : usual care of in a medico-social service (medical, social, neuropsychological and psychological),
  2. 5 months of dialectical behavior therapy (DBT)
     -DBT skills training group : during 19 weeks
  3. 5 months of follow-up : usual care of + monthly reminders of DBT intervention skills
  Interventions: Behavioral: Dialectical Behavior Therapy and Radically Open dialectical behavior therapy
- Controls without brain injury (No Intervention): People without brain injury used as controls for linguistic markers of emotional expression regulation and free will.
- GREMO patients' family (No Intervention): GREMO patients' relatives, without brain injury, living with the GREMO patient and ready to complete every day and adapted self-observational diary card similar to the one of the GREMO patient
- Qualitative research ABI patients and families (No Intervention): Patients and relatives followed by the same medico-social service but not meeting GREMO patients eligibility criteria, participating only in the qualitative research on free will and spirituality

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy and Radically Open dialectical behavior therapy — Dialectical Behavior Therapy is a third wave cognitive-behavioral therapy. It focuses on emotional dysregulation and interactions between the patient and his family in genesis and maintenance of challenging behaviors. It is used here in an adapted form for cognitive problems.
  Delivered in a group format of 19 weeks + individual sessions.
  Arms: GREMO patients

SUMMARY:
After acquired brain injury (ABI), persons can experience emotional and behavioral difficulties, that can be painful both for the person and his/her family. This clinical study aims at measuring the effectiveness of a third wave cognitive behavioral therapy called "dialectical behavior therapy" (DBT). DBT aims at teaching persons emotion regulation skills, interpersonal effectiveness skills, mindfulness and distress tolerance skills through group and individual sessions.

The study's hypothesis is that DBT, in an adapted format for persons with ABI can lead to

* a better quality of life, emotional and behavioral regulation, and self-esteem
* decrease in problematic behaviors
* progress in life goals
* increase post traumatic growth and spirituality
* better family functioning and lesser burden for care givers
* experiencing more emotions and more free will

  45 persons with an ABI sustained more than 18 month back, will follow a 3 phases, follow-up with care as usual for 5 months, followed by 5 months of DBT, followed by 5 months of care as usual + DBT monthly sessions.

Self- and family-questionnaire will explore quality of life, emotional regulation, self-esteem, stress, anxiety, cognitive difficulties, family functioning and coping, post traumatic growth and spirituality and will be compared across the 3 phases. Results will be analyzed at a group level but also at an individual level (each patient separately) to test for decrease in unwanted behaviors and at a dyadic level (the person and his/her spouse) to test for the mutual effect of regulating emotions. Persons' memories will by analyzed at 3 time points by a linguistic analysis, and experience of free will after ABI will be analyzed by transcribed narratives of participants.

DETAILED DESCRIPTION:
The study will explore the impact of Dialectical Behavior Therapy (DBT) skills training on patients with ABI, their families and on for their family system interactions.

->Triple methodology :

1. 3 stages, monocentric, comparative, open-label for part of the outcome measures and single-blinded (only for linguistic markers) with active control treatment
2. Prospective (at the individual level) and correlational (at the dyad level: client - family member) single-case experimental study exploring emotional-behavioral interactions as a function of the use of DBT skills by the client, over time.

   Further, it will explore the experience of free will (the property of the human will to determine itself freely), in relation to emotions and meaning of life/spirituality after ABI and the modifications of this experience after DBT.
3. qualitative study of semi-structured individual by Interpretative Phenomenological Analysis (IPA

The objectives of this research are to show that a group training of DBT skills allows persons with ABI, (1) to improve quality of life - main objective; (2) to improve self-esteem and emotional regulation (3) to decrease depressive symptoms and problematic behaviors, (4) to self-determine and achieve one's goals (Goal Attainment Scaling) for a life worth living; (5) to improve coping and family functioning; (7) to decrease caregiver burden; (8) to interpret one's life, with more expression of emotions, non-judgment, acceptance of the difficulty of life and motivation to change (measured by linguistic analysis of emotionally charged memories)

ELIGIBILITY:
Eligibility Criteria: * (Limit: 15,000 characters)

Summary criteria for participant selection.

Main eligibility criteria

GREMO patients :

* Inclusion criteria:

  * Persons with acquired brain injury regardless of the type or location of the injury
  * Age between 18 and 68
  * Over 18 months since the acquired brain injury (or 6 month if mild traumatic brain injury)
  * Challenging behaviors or emotional dysregulation or high level of anxiety / depression or family's complaints about emotional dysregulation
  * Secondary or exacerbated by an acquired brain injury
  * Causing important suffering for themselves or their families
  * Being affiliated to a social security
  * Fluent in French
  * Being able to understand goals and risks and to give a dated and signed consent
* Exclusion criteria:

  * Clinically evident severe lack of insight, lack of abstract reasoning, or severe anosognosia
  * Patients without any complaints
  * Severe cognitive impairments, aphasia or intellectual impairments that doesn't allow to understand DBT skills, questionnaires or group intreactions
  * Non fluent in French
  * Associated brain degenerative disease
  * Cancerous brain injury with uncertain progression
  * Non-stabilized psychotic disorder
  * Following a third wave cognitive behavioral therapy during the research study (for example : acceptance and commitment therapy)

Controls without brain injury

* Inclusion criteria :

  * Being 18 years old or more
  * Without brain injury
* Exclusion criteria :

  * Non fluent in French
  * History of brain injury or brain disease
  * History of psychiatric disorder
  * Personality disorder
  * GREMO patient's family member living together
  * Psychologist, neuropsychologist or people with an emotional regulation knowledge linked to their profession
  * Being under guardianship or curatorship
  * Being pregnant or breastfeeding

GREMO patients' family members

* Inclusion criteria :

  * Being 18 years old or more
  * GREMO patient's family member
  * Living with a GREMO patient
  * Agreeing to rate an emotion-behavior-skills diary cards
* Exclusion criteria :

  * GREMO patient's refusal for their family member to participate
  * Non fluent in French
  * Brain injury or brain disease
  * Major lack of insight
  * Being under trusteeship or curatorship

Qualitative research ABI patients and families

* Inclusion criteria :

  * Person with ABI attending the same medico-social service as GREMO patients
  * Ineligible for GREMO patients group (participation refusal, major insight difficulty…)
  * Agreeing to talk about their free will or spirituality
* Exclusion criteria :

  * Aphasia or dysarthria not allowing understandable recording
  * Impossibility to understand oral questions
  * Non fluent in French

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Quality Of Life after Brain Injury | 15 months
  Evaluation of quality of life after brain injury with QOLIBRI (Quality Of Life after Brain Injury)on 37 items belonging to 6 factors: cognition, self, daily life and autonomy, social relationships, emotions and physical problems. The Qolibri scores are reported a 0-100. 0 is the worst and 100 is the best.
  Self-rated by GREMO patients.

SECONDARY OUTCOMES:
Evaluation of the difficulties in emotions regulation | 15 months
  Evaluation of emotional regulation difficulties with DERS ( Difficuties en Emotion Regulation Scale)-16 on 16 items filed in 5 factors : lack of emotional clarity, difficulties engaging in goal-directed behavior, impulse control difficulties, limited access to effective emotion regulation strategies, nonacceptance of emotional responses.
  Self-rated by GREMO patients and self-rated by family member about themselves. DERS-16 can range from 16 to 80, higher scores suggest greater problems with emotion regulation
Evaluation of self-esteem | 15 months
  Evaluation of self-esteem on 10 items with EES-10 (Rosenberg Self-Esteem Scale) . You then get a score between 10 and 40.If you score below 25, your self-esteem is very low. Work in this area seems desirable. If you get a score above 39, your self-esteem is very high and you tend to be strongly assertive.
  Self-rated by GREMO patients
Evaluation of executive functioning | 15 months
  Evaluation of executive functioning with BRIEF-A (Behavior Rating Inventory of Executive Function-Adult Version) on 75 items filed in inhibit, self-monitor, plan/organize, shift, initiate, task monitor, emotional control, working memory and organization of materials.
  Self-rated by GREMO patients and proxi-rated by a family member.high scores obtained on the BRIEF do not indicate a "disorder of executive function" but rather suggest a higher level of dysfunction in a specific domain of executive functions
Evaluation of reflective functioning | 15 months
  Evaluation of reflective functioning with RFQ (Reflective Function Questionnaire) on 8 items.
  7 if you strongly agree, and the 1 if you arestrongly disagree. Use the middle point (the 4) if you are neutral or indecisive requirements of the RFQ
Evaluation of psychological distress | 15 months
  Evaluation of psychological distress with DASS-21 (Depression Anxiety Stress Scale) on 21 items about depression, anxiety and stress.
  Each of the 21 questions is scored on a 4-point scale ranging from 0 ("Did not apply to me at all") to 3 ("Applied to me very much, or most of the time"). Scores for Depression,
  Anxiety and Stress are calculated by summing the scores for the relevant items:
  Depression: 3, 5, 10, 13, 16, 17, 21 Anxiety: 2, 4, 7, 9, 15, 19, 20 Stress: 1, 6, 8, 11, 12, 14, 1
Evaluation of positive outcomes reported by persons who have experienced traumatic event | 15 months
  Evaluation of positive outcomes reported by persons who have experienced traumatic events, such as brain injury, which evaluates new possibilities, relating to others, personal strength, spiritual change, and appreciation of life with Post-traumatic Growth Inventory.
  Self-rated by GREMO patients. It consists of 21 questions to which responses are given on a scale of 0-5, with 0 representing no change and 5 showing a great degree of change.
Evaluation of the perception of the family functioning | 15 months
  Evaluation of the perception of the family functioning on 12 items with FAD (Family Assessment Device). Scores range from 1 to 4 with 1 reflecting healthy functioning and 4 reflecting unhealthy functioning.
Evaluation of coping cope with dysfunctions related to their relatives' pathology. | 15 months
  Evaluation of coping cope with dysfunctions related to their relatives' pathology.
  Rated by a family member with FCQ (Family Coping Questionnaire).It consists of 21 questions to which responses are given on a scale of 0-5, with 0 representing no change and 5 showing a great degree of change.
Evaluation of family burden | 15 months
  Evaluation of family burdenon 21 items with Zarit (Zarit Burden Interview) questionnaire
  Rated by a family member.The Zarit Burden Interview (ZBI) The ZBI consists of 22 items rated on a 5-point Likert scale that ranges from 0 (never) to 4 (nearly always) with the sum of scores ranging between 0-88. Higher scores indicate greater burden. A score of 17 or more was considered high burden
Evaluation of the goal attainment related to better emotional regulation | 15 months
  3 milestone, 5-level GAS, evaluating goal attainment related to better emotional regulation. Each GREMO patient will have at least on personalized GAS according to his/her goals with Goal Attainment Scaling.
  0 means not important, 1 means important, 2 means very important and 3 means extremely important

CONTACTS AND LOCATIONS:
Locations (1):
- Service EMOI-TC - Pôle de MPR Institut Universitaire de Réadaptation Clemenceau (IURC), Illkirch-Graffenstaden, France

IPD SHARING:
Plan to Share IPD: Undecided